CLINICAL TRIAL: NCT00814749
Title: a Multicentered Randomised Controlled Trial to Test the Cost Effectiveness of Urodynamics in Women With Symptoms of Stress Urinary Incontinence in Whom Surgical Treatment is Considered
Brief Title: Value of Urodynamics Prior to Stress Incontinence Surgery 2
Acronym: VUSIS 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006/197
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Last update posted 2008-12-25 (Estimated); Status verified 2008-12

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; urodynamics; randomized clinical trial; surgery
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgical therapy (Active Comparator)
  Interventions: Procedure: midureteral sling
- individual management (Active Comparator)
  Interventions: Other: surgical therapy or conservative

INTERVENTIONS:
Procedure: midureteral sling — midureteral sling
  Arms: surgical therapy
Other: surgical therapy or conservative — midureteral sling or conservative; medication, physiotherapy
  Arms: individual management

SUMMARY:
To test the value of preoperatively performed urodynamics with regard to outcome of surgery for stress urinary incontinence (SUI) and to examine whether not performing urodynamics preoperatively is more cost effective than performing urodynamics preoperatively using the non-inferiority assumption.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of stress urinary incontinence and/or mixed urinary incontinence, predominantly stress incontinence
* Signs of stress urinary incontinence on physical examination or voiding-diary
* Patient is a candidate for surgical treatment (as based on history and physical examination)
* Patient has attended at least 3 months of physiotherapy
* Patient accepts randomisation
* Patient is capable to fill out bladder diary's, pad tests and questionnaires
* Patient understands the Dutch written and spoken language
* ASA 1 or 2

Exclusion Criteria:

* Previous incontinence surgery
* Mixed urinary incontinence, urge component is predominant
* Prolapse >= 1cm beyond the hymen on Valsalva in supine position
* Postvoid urinary residual > 150ml
* Present urinary tract infection
* The need for additional pelvic surgery (prolapse and/or hysterectomy)
* Patient is or wants to become pregnant
* Prior pelvic radiotherapy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Non inferiority of the improvement of the urinary distress inventory one year after treatment. | one year

SECONDARY OUTCOMES:
Cure of incontinence as measured with voiding diary. Complications of surgery for stress urinary incontinence, in particular re-operations and overactive bladder symptoms. Quality of life as measured by RAND-36, Euroqol and IIQ. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Vierhout, MD, PhD, Principal Investigator — Radboud University Medical Center; John Heesakkers, MD, PhD, Principal Investigator — University Medical Center St. Radboud; Kirsten Kluivers, MD, PhD, Principal Investigator — University Medical Center St. Radboud; Sanne van Leijsen, MD, Principal Investigator — University Medical Center St. Radboud; Ben Willem Mol, MD, PhD, Principal Investigator — Academic Medical Centre Amsterdam
Locations (1):
- University Medical Center St. Radboud, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] van Leijsen SAL, Kluivers KB, Mol BWJ, Hout J', Milani AL, Roovers JWR, Boon JD, Vaart CHV, Langen PH, Hartog FE, Dietz V, Tiersma ESM, Hovius MC, Bongers MY, Spaans W, Heesakkers JPFA, Vierhout ME; Dutch Urogynecology Consortium*. Value of urodynamics before stress urinary incontinence surgery: a randomized controlled trial. Obstet Gynecol. 2013 May;121(5):999-1008. doi: 10.1097/AOG.0b013e31828c68e3. PMID 23635736
- [Derived] van Leijsen SA, Kluivers KB, Mol BW, Broekhuis SR, Milani FL, van der Vaart CH, Roovers JP, Bongers MY, den Boon J, Spaans WA, de Leeuw JW, Dietz V, Kleinjan JH, Brolmann HA, Roos EJ, Schaafstra J, Heesakkers JP, Vierhout ME. Protocol for the value of urodynamics prior to stress incontinence surgery (VUSIS) study: a multicenter randomized controlled trial to assess the cost effectiveness of urodynamics in women with symptoms of stress urinary incontinence in whom surgical treatment is considered. BMC Womens Health. 2009 Jul 21;9:22. doi: 10.1186/1472-6874-9-22. PMID 19622153